CLINICAL TRIAL: NCT01260038
Title: Personalized 1st-line Treatment of Patients With NSCLC: is Timely Analysis of EGFR-mutation Status Feasible in a Routine Practice Setting in Antwerp.
Brief Title: Study in NSCLC: is Timely Analysis of EGFR-mutation Status Feasible in Region Antwerp, Belgium.
Acronym: HERMES
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); AstraZeneca (Industry)
Responsible Party: Thoracale Oncologie Groep Antwerpen, Universiteit Antwerpen
Other Study IDs: TOGA 1001
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; observational study; EGFR mutation analysis; EGFR mutation status; testing turn around time
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — At diagnosis a tumor sample is collected for histological evaluation, this sample will be used for the biomarker analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to evaluate the feasibility of the implementation of a personalized treatment strategy based on specific tumor marker (f.i. EGFR-mutation) in the routine clinical care setting in the Antwerp region (Belgium).

DETAILED DESCRIPTION:
The favourable results of a number of phase III-trials with gefitinib in NSCLC patients with activating EGFR-mutations, have resulted in the licensing of gefitinib in this indication. This offers the prospect of a true personalized treatment of patients with NSCLC. Implementation of such a personalized treatment strategy is dependent both on the availability of adequate tumor samples for the EGFR-mutation analysis and on the timely reporting of the mutation analysis results. Ideally the results should be available in all patients within 2 weeks of the analysis request.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* newly diagnosed NSCLC
* written informed consent
* tumor sample available

Exclusion Criteria:

* mixed histology of small cell and NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed patients with Non Small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
testing turn around time (in days) | up to 1 month
  how long does it take to get the mutation analysis result

SECONDARY OUTCOMES:
demographics | baseline
  age, gender, tumor histology, smoking history
correlation between pulmonary function/pulmonary antecedents and EGFR-mutation status | baseline
correlation between family history with regards to cancer and EGFR-mutation status | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Germonpre, MD, Principal Investigator — UZA + Thoracale Oncologie Groep Antwerpen
Locations (11):
- Belgium (11):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - AZ Monica, Antwerp
  - GZA Sint Vincentius - Sint Augustinus, Antwerp
  - ZNA Middelheim - ZNA STER - ZNA Jan Palfijn, Antwerp
  - AZ St Jozef Bornem en Willebroek, Bornem
  - AZ Klina, Brasschaat
  - AZ St Dimpna, Geel
  - AZ St Elisabeth, Herentals
  - AZ Mol, Mol
  - AZ Nikolaas, Sint-Niklaas
  - AZ Turnhout, Turnhout